CLINICAL TRIAL: NCT02452190
Title: A 52-Week Double-Blind, Placebo-Controlled, Parallel-Group Efficacy and Safety Study of Reslizumab 110 mg Fixed, Subcutaneous Dosing in Patients With Uncontrolled Asthma and Elevated Blood Eosinophils
Brief Title: Study of Reslizumab in Participants With Uncontrolled Asthma and Elevated Blood Eosinophils
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C38072-AS-30025; 2015-000865-29 (EudraCT Number)
Record Dates: First submitted 2015-05-13; First posted 2015-05-22 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — reslizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reslizumab (Experimental): Reslizumab
  Interventions: Drug: Reslizumab
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reslizumab — Reslizumab will be administered subcutaneously in a dose of 110 mg every 4 weeks.
  Arms: Reslizumab
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the effect of reslizumab (110 mg) administered subcutaneously every 4 weeks on clinical asthma exacerbations in adults and adolescents with asthma and elevated blood eosinophils who are inadequately controlled on standard-of-care asthma therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained.
* The participant is male or female, 12 years of age and older, with a diagnosis of asthma.
* The participant has Forced Expiratory Volume in 1 Second (FEV1) reversibility according to standard American Thoracic Society (ATS) or European Respiratory Society (ERS) protocol.
* The participant has required an inhaled corticosteroid.
* The participant has required an additional asthma controller medication besides inhaled corticosteroids.
* The participant has a history of asthma exacerbation.
* The participant must be willing and able to comply with study restrictions, perform requisite procedures and remain at the clinic for the required duration during the study period, and be willing to return to the clinic for the follow-up evaluation as specified in this protocol.

  * Additional criteria may apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has any clinically significant, uncontrolled medical condition (treated or untreated) that would interfere with the study schedule or procedures, interpretation of efficacy results, or compromise the patient's safety.
* The participant has another confounding underlying lung disorder
* The participant has a known hypereosinophilic syndrome.
* The participant has a diagnosis of malignancy within 5 years of the screening visit, except for treated and cured non-melanoma skin cancers.
* The participant is a pregnant or lactating woman, or intends to become pregnant during the study. Any woman becoming pregnant during the study will be withdrawn from the study.
* The participant is a current smoker or has a smoking history.
* The participated in a clinical trial within 30 days or 5 half-lives of the investigational drug before screening, whichever is longer.
* The participant was previously exposed to reslizumab.
* The participant has a history of an immunodeficiency disorder including human immunodeficiency virus (HIV).
* The participant has current or suspected drug and alcohol abuse.
* The participant has an active helminthic parasitic infection or was treated for one within 6 months of screening.
* The participant has a history of allergic reaction or hypersensitivity to any component of the study drug.

  * Additional criteria may apply, please contact the investigator for more information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (226):
- United States (69):
  - Teva Investigational Site 13212, Birmingham, Alabama
  - Teva Investigational Site 13241, Flagstaff, Arizona
  - Teva Investigational Site 13194, Glendale, Arkansas
  - Teva Investigational Site 13215, Bakersfield, California
  - Teva Investigational Site 13181, Canoga Park, California
  - Teva Investigational Site 13254, Fresno, California
  - Teva Investigational Site 13216, Huntington Beach, California
  - Teva Investigational Site 13247, Long Beach, California
  - Teva Investigational Site 13205, Napa, California
  - Teva Investigational Site 13764, San Jose, California
  - Teva Investigational Site 13252, Stockton, California
  - Teva Investigational Site 13251, Walnut Creek, California
  - Teva Investigational Site 13229, Denver, Colorado
  - Teva Investigational Site 13766, Waterbury, Connecticut
  - Teva Investigational Site 13196, Aventura, Florida
  - Teva Investigational Site 13256, Fort Lauderdale, Florida
  - Teva Investigational Site 13203, Kissimmee, Florida
  - Teva Investigational Site 13197, Miami, Florida
  - Teva Investigational Site 13220, Miami, Florida
  - Teva Investigational Site 13243, Miami, Florida
  - Teva Investigational Site 13233, New Port Richey, Florida
  - Teva Investigational Site 13201, Orlando, Florida
  - Teva Investigational Site 13250, Orlando, Florida
  - Teva Investigational Site 13246, Pembroke Pines, Florida
  - Teva Investigational Site 13208, Tallahassee, Florida
  - Teva Investigational Site 13255, Tampa, Florida
  - Teva Investigational Site 13765, Albany, Georgia
  - Teva Investigational Site 13249, Buford, Georgia
  - Teva Investigational Site 13763, Lawrenceville, Georgia
  - Teva Investigational Site 13230, Chicago, Illinois
  - Teva Investigational Site 13211, Normal, Illinois
  - Teva Investigational Site 13235, Shiloh, Illinois
  - Teva Investigational Site 13202, Michigan City, Indiana
  - Teva Investigational Site 13225, Lenexa, Kansas
  - Teva Investigational Site 13222, Owensboro, Kentucky
  - Teva Investigational Site 13191, Lafayette, Louisiana
  - Teva Investigational Site 13200, North Dartmouth, Massachusetts
  - Teva Investigational Site 13226, Biloxi, Mississippi
  - Teva Investigational Site 13204, St Louis, Missouri
  - Teva Investigational Site 13258, Boys Town, Nebraska
  - Teva Investigational Site 13769, Belleville, New Jersey
  - Teva Investigational Site 13210, Ocean City, New Jersey
  - Teva Investigational Site 13188, New Hyde Park, New York
  - Teva Investigational Site 13232, New York, New York
  - Teva Investigational Site 13767, New York, New York
  - Teva Investigational Site 13186, Cincinnati, Ohio
  - Teva Investigational Site 13253, Cleveland, Ohio
  - Teva Investigational Site 13240, Toledo, Ohio
  - Teva Investigational Site 13259, Edmond, Oklahoma
  - Teva Investigational Site 13238, Oklahoma City, Oklahoma
  - Teva Investigational Site 13195, Medford, Oregon
  - Teva Investigational Site 13242, Bethlehem, Pennsylvania
  - Teva Investigational Site 13218, Jenkintown, Pennsylvania
  - Teva Investigational Site 13189, Philadelphia, Pennsylvania
  - Teva Investigational Site 13190, Pittsburgh, Pennsylvania
  - Teva Investigational Site 13209, East Providence, Rhode Island
  - Teva Investigational Site 13217, Lincoln, Rhode Island
  - Teva Investigational Site 13223, Knoxville, Tennessee
  - Teva Investigational Site 13185, Arlington, Texas
  - Teva Investigational Site 13199, Corsicana, Texas
  - Teva Investigational Site 13260, Dallas, Texas
  - Teva Investigational Site 13224, San Antonio, Texas
  - Teva Investigational Site 13184, Waco, Texas
  - Teva Investigational Site 13187, Provo, Utah
  - Teva Investigational Site 13207, Abingdon, Virginia
  - Teva Investigational Site 13183, Fairfax, Virginia
  - Teva Investigational Site 13257, Falls Church, Virginia
  - Teva Investigational Site 13239, Richmond, Virginia
  - Teva Investigational Site 13227, Spokane, Washington
- Argentina (11):
  - Teva Investigational Site 20040, Buenos Aires
  - Teva Investigational Site 20033, Buenos Aires
  - Teva Investigational Site 20035, Buenos Aires
  - Teva Investigational Site 20041, Córdoba
  - Teva Investigational Site 20053, Lanús
  - Teva Investigational Site 20037, Mar del Plata
  - Teva Investigational Site 20036, Mendoza
  - Teva Investigational Site 20054, Rosario
  - Teva Investigational Site 20032, Rosario
  - Teva Investigational Site 20046, San Miguel de Tucumán
  - Teva Investigational Site 20045, San Rafael
- Australia (5):
  - Teva Investigational Site 78085, Bedford Park
  - Teva Investigational Site 78083, Nedlands
  - Teva Investigational Site 78088, Parkville
  - Teva Investigational Site 78087, Sherwood
  - Teva Investigational Site 78084, Woolloongabba
- Belgium (3):
  - Teva Investigational Site 37054, Brussels
  - Teva Investigational Site 37053, Erpent
  - Teva Investigational Site 37055, Ghent
- Canada (3):
  - Teva Investigational Site 11106, Vancouver, British Columbia
  - Teva Investigational Site 11105, Etobicoke, Ontario
  - Teva Investigational Site 11109, Windsor
- Czechia (3):
  - Teva Investigational Site 54130, Jablonec nad Nisou
  - Teva Investigational Site 54128, Jindřichův Hradec
  - Teva Investigational Site 54129, Tábor
- France (2):
  - Teva Investigational Site 35182, Strasbourg
  - Teva Investigational Site 35183, Toulouse
- Germany (16):
  - Teva Investigational Site 32559, Bad Wörishofen
  - Teva Investigational Site 32556, Berlin
  - Teva Investigational Site 32561, Berlin
  - Teva Investigational Site 32570, Berlin
  - Teva Investigational Site 32567, Berlin
  - Teva Investigational Site 32564, Berlin
  - Teva Investigational Site 32568, Frankfurt
  - Teva Investigational Site 32560, Frankfurt am Main
  - Teva Investigational Site 32562, Hamburg
  - Teva Investigational Site 32566, Hanover
  - Teva Investigational Site 32555, Koblenz
  - Teva Investigational Site 32563, Leipzig
  - Teva Investigational Site 32557, Leipzig
  - Teva Investigational Site 32565, Lübeck
  - Teva Investigational Site 32551, Mainz
  - Teva Investigational Site 32569, Witten
- Hungary (16):
  - Teva Investigational Site 51216, Balassagyarmat
  - Teva Investigational Site 51228, Budapest
  - Teva Investigational Site 51221, Csorna
  - Teva Investigational Site 51220, Debrecen
  - Teva Investigational Site 51223, Debrecen
  - Teva Investigational Site 51255, Dombóvár
  - Teva Investigational Site 51218, Gödöllő
  - Teva Investigational Site 51222, Győr
  - Teva Investigational Site 51227, Hajdúnánás
  - Teva Investigational Site 51226, Kaposvár
  - Teva Investigational Site 51231, Kapuvár
  - Teva Investigational Site 51224, Százhalombatta
  - Teva Investigational Site 51219, Szeged
  - Teva Investigational Site 51225, Szigetvár
  - Teva Investigational Site 51217, Szombathely
  - Teva Investigational Site 51229, Veszprém
- Israel (9):
  - Teva Investigational Site 80077, Ashkelon
  - Teva Investigational Site 80076, Haifa
  - Teva Investigational Site 80094, Jerusalem
  - Teva Investigational Site 80078, Jerusalem
  - Teva Investigational Site 80080, Kfar Saba
  - Teva Investigational Site 80073, Petah Tikva
  - Teva Investigational Site 80081, Petah Tikva
  - Teva Investigational Site 80079, Ramat Gan
  - Teva Investigational Site 80075, Rehovot
- Japan (18):
  - Teva Investigational Site 84039, Amagasaki
  - Teva Investigational Site 84053, Ginowan
  - Teva Investigational Site 84049, Hakodate
  - Teva Investigational Site 84034, Hiroshima
  - Teva Investigational Site 84036, Kanazawa
  - Teva Investigational Site 84037, Kishiwada-shi
  - Teva Investigational Site 84048, Kobe
  - Teva Investigational Site 84044, Kobe
  - Teva Investigational Site 84047, Kodaira
  - Teva Investigational Site 84045, Kumamoto
  - Teva Investigational Site 84043, Mizunami-shi
  - Teva Investigational Site 84041, Sagamihara
  - Teva Investigational Site 84031, Tokyo
  - Teva Investigational Site 84032, Tokyo
  - Teva Investigational Site 84038, Toyama
  - Teva Investigational Site 84046, Toyama
  - Teva Investigational Site 84035, Toyoake-shi
  - Teva Investigational Site 84040, Yokohama
- Mexico (6):
  - Teva Investigational Site 21084, Guadalajara
  - Teva Investigational Site 21085, Guadalajara
  - Teva Investigational Site 21088, Guadalajara
  - Teva Investigational Site 21089, Guadalajara
  - Teva Investigational Site 21087, Monterrey
  - Teva Investigational Site 21086, Zapopan
- New Zealand (2):
  - Teva Investigational Site 79047, Auckland
  - Teva Investigational Site 79046, Auckland
- Poland (8):
  - Teva Investigational Site 53310, Bialystok
  - Teva Investigational Site 53315, Bialystok
  - Teva Investigational Site 53308, Gdansk
  - Teva Investigational Site 53311, Krakow
  - Teva Investigational Site 53314, Lodz
  - Teva Investigational Site 53312, Lodz
  - Teva Investigational Site 53313, Poznan
  - Teva Investigational Site 53309, Tarnów
- Romania (8):
  - Teva Investigational Site 52108, Brasov
  - Teva Investigational Site 52109, Brasov
  - Teva Investigational Site 52107, Bucharest
  - Teva Investigational Site 52105, Bucharest
  - Teva Investigational Site 52104, Cluj-Napoca
  - Teva Investigational Site 52111, Deva
  - Teva Investigational Site 52106, Târgu Mureş
  - Teva Investigational Site 52110, Timișoara
- Russia (8):
  - Teva Investigational Site 50350, Barnaul
  - Teva Investigational Site 50354, Kemerovo
  - Teva Investigational Site 50348, Moscow
  - Teva Investigational Site 50351, Moscow
  - Teva Investigational Site 50347, Novosibirsk
  - Teva Investigational Site 50355, Saint Petersburg
  - Teva Investigational Site 50352, Saint Petersburg
  - Teva Investigational Site 50349, Tomsk
- South Africa (7):
  - Teva Investigational Site 90027, Benoni
  - Teva Investigational Site 90028, Bloemfontein
  - Teva Investigational Site 90026, Cape Town
  - Teva Investigational Site 90031, Cape Town
  - Teva Investigational Site 90029, Cape Town
  - Teva Investigational Site 90032, Durban
  - Teva Investigational Site 90030, Durban
- South Korea (3):
  - Teva Investigational Site 87015, Bucheon-si
  - Teva Investigational Site 87016, Seoul
  - Teva Investigational Site 87014, Seoul
- Spain (4):
  - Teva Investigational Site 31149, Barcelona
  - Teva Investigational Site 31147, Esplugues de Llobregat
  - Teva Investigational Site 31152, Girona
  - Teva Investigational Site 31154, Vitoria-Gasteiz
- Turkey (Türkiye) (5):
  - Teva Investigational Site 82042, Ankara
  - Teva Investigational Site 82041, Izmir
  - Teva Investigational Site 82040, Kocaeli
  - Teva Investigational Site 82039, Konya
  - Teva Investigational Site 82043, Mersin
- Ukraine (20):
  - Teva Investigational Site 58216, Chernivtsi
  - Teva Investigational Site 58219, Dnipropetrovsk
  - Teva Investigational Site 58225, Dnipropetrovsk
  - Teva Investigational Site 58222, Ivano-Frankivsk
  - Teva Investigational Site 58227, Kharkiv
  - Teva Investigational Site 58213, Kharkiv
  - Teva Investigational Site 58221, Kharkiv
  - Teva Investigational Site 58223, Kharkiv
  - Teva Investigational Site 58214, Kremenchuk
  - Teva Investigational Site 58228, Kryvyi Rih
  - Teva Investigational Site 58220, Kyiv
  - Teva Investigational Site 58230, Kyiv
  - Teva Investigational Site 58218, Kyiv
  - Teva Investigational Site 58226, Kyiv
  - Teva Investigational Site 58253, Kyiv
  - Teva Investigational Site 58234, Sumy
  - Teva Investigational Site 58229, Vinnytsia
  - Teva Investigational Site 58233, Vinnytsia
  - Teva Investigational Site 58231, Zaporizhzhya
  - Teva Investigational Site 58224, Zhaporizhzhya

REFERENCES:
- [Derived] Bernstein JA, Virchow JC, Murphy K, Maspero JF, Jacobs J, Adir Y, Humbert M, Castro M, Marsteller DA, McElhattan J, Hickey L, Garin M, Vanlandingham R, Brusselle G. Effect of fixed-dose subcutaneous reslizumab on asthma exacerbations in patients with severe uncontrolled asthma and corticosteroid sparing in patients with oral corticosteroid-dependent asthma: results from two phase 3, randomised, double-blind, placebo-controlled trials. Lancet Respir Med. 2020 May;8(5):461-474. doi: 10.1016/S2213-2600(19)30372-8. Epub 2020 Feb 14. PMID 32066536

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1159 participants were screened, of whom 468 participants were eligible and enrolled in a 3-week run-in period for self-monitoring. All 468 enrolled participants were then randomized at 201 centers in 20 countries.
Groups:
- Placebo: Matching placebo administered subcutaneously once every 4 weeks (+/-7 days) for a total of 13 doses.
- Reslizumab 110 mg: Reslizumab 110 milligrams (mg) administered subcutaneously once every 4 weeks (+/-7 days) for a total of 13 doses.
Period: Overall Study
Arm/Group | Placebo | Reslizumab 110 mg
Started | 232 | 236
Intent to Treat (ITT) Population (All randomized participants, excluding 4 from a terminated study site.) | 230 | 234
Safety Population (Placebo participant treated with reslizumab at 1 visit is counted in reslizumab arm for Safety.) | 231 | 237
Completed | 197 | 212
Not Completed | 35 | 24
Not completed — Withdrawal by Sponsor | 1 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Investigator's Decision | 2 | 0
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 4 | 3
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 20 | 11
Not completed — Noncompliance with study drug | 1 | 0
Not completed — Participant traveled abroad | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population includes all randomized participants, excluding participants from the site terminated due to Good Clinical Practice (GCP) issues. Treatment was based on the treatment to which participants were randomized, regardless of which treatment they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Reslizumab 110 mg | Total
Number analyzed (Participants) | 230 | 234 | 464
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (17.70) | 46.9 (17.63) | 45.9 (17.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 144 | 272
  Male | 102 | 90 | 192
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 201 | 216 | 417
  Hispanic or Latino | 26 | 17 | 43
  Unknown | 3 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 199 | 205 | 404
  Black or African American | 11 | 15 | 26
  Asian | 11 | 6 | 17
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 8 | 8 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States and Canada | 58 | 52 | 110
  Europe | 125 | 135 | 260
  Rest of World | 47 | 47 | 94
Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] — Population: Participants in the ITT population with re-bronchodilator FEV1 at baseline measures available.
  liters
    number analyzed (Participants) | 229 | 234 | 463
    (all) | 2.102 (0.870) | 1.988 (0.780) | 2.044 (0.827)
Asthma Quality of Life Questionnaire for Participants 12 Years and Older (AQLQ+12) Score [Mean (Standard Deviation); unit: units on a scale] — AQLQ is a 32-item instrument administered as a self-assessment. AQLQ+12 is a modified version of AQLQ developed to measure functional impairments of participants aged 12-70 years. It is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Participants were asked to recall their experiences during the last 2 weeks and respond to each question on a 7-point scale (1=severe impairment, 7=no impairment), where higher scores indicated "better quality of life." Overall AQLQ+12 score is the mean of all 32 responses. Population: Participants in the ITT population with baseline AQLQ+12 scores available
  units on a scale
    number analyzed (Participants) | 215 | 217 | 432
    (all) | 4.39 (0.995) | 4.28 (1.048) | 4.33 (1.022)
Asthma Control Questionnaire (ACQ-6) Score [Mean (Standard Deviation); unit: units on a scale] — The ACQ-6 is a validated 6-item asthma assessment tool that has been widely used. Six questions are self-assessments (completed by the participant), 5 questions assessing asthma symptoms: night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and 1 question for short-acting bronchodilator use. Each item on the ACQ has a possible score ranging from 0 to 6, and the total score is the mean of all responses. The total score ranging from 0-6 (0=totally controlled and 6=severely uncontrolled).
  units on a scale | 2.42 (0.812) | 2.48 (0.88) | 2.45 (0.847)
Total Asthma Symptom Scores [Mean (Standard Deviation); unit: units on a scale] — Asthma symptoms were recorded by participants in an asthma control diary. Night score was assessed on a 5-point scale where 0=no symptoms, slept through night, to 4=bad night, no sleep. Day score was assessed on a 6-point scale where 0=very well, no symptoms, to 5=asthma very severe, unable to carry out daily activities. Total asthma symptom score was calculated by taking the sum of the night and day asthma symptom scores recorded each day, ranging from 0 (no symptom) to 9 (severe symptom). Population: Participants in the ITT population with total asthma symptom scores at baseline.
  units on a scale
    number analyzed (Participants) | 222 | 224 | 446
    (all) | 2.6 (1.62) | 2.5 (1.53) | 2.57 (1.578)
Blood Eosinophil Category at Baseline [Count of Participants; unit: Participants] — Population: Participants with eosinophil count at baseline stratification data available.
  Participants
    less than (<)300 per (/) microliter (µL) | 0 | 1 | 1
    300 to <400/µL | 42 | 48 | 90
    greater than or equal to (≥)400/µL | 188 | 185 | 373
Number of Clinical Asthma Exacerbation (CAE) Events in the Previous 12 Months [Mean (Standard Deviation); unit: Count of Events] — CAE was defined at baseline as asthma exacerbations requiring systemic corticosteroids within last 12 months.
  Count of Events | 2.30 (0.843) | 2.35 (1.043) | 2.33 (0.949)

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinical Asthma Exacerbations (CAEs) During 52 Weeks of Treatment
Description: A CAE was defined as a clinically-judged deterioration in asthma control, as determined by the investigator and as evidenced by new or worsening asthma signs or symptoms based on the participant's history, asthma control diary, physical examination, and/or ambulatory or clinic visit assessment of lung function and that resulted in a medical intervention, including at least 1 of the following: 1) use of systemic corticosteroids (oral or injection) or at least a doubling from a stable maintenance oral corticosteroid dose for at least 3 days; 2) asthma-specific hospital admission; 3) asthma-specific emergency department visit. Adjusted CAE rate and confidence intervals were based on Negative Binomial regression model adjusted for stratification factors. Results are presented as adjusted means. For this analysis, the offset variable is calculated as the logarithm of treatment duration minus the summed duration of exacerbations during the treatment period.
Time Frame: Day 1 to Week 52
Population: ITT population included all randomized participants, excluding participants from the site terminated due to GCP issues. Treatment was based on the treatment to which participants were randomized, regardless of which treatment they received.
Measure: Mean (95% Confidence Interval); unit: events
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 230 | 234
events | 0.52 [0.347 to 0.773] | 0.41 [0.279 to 0.607]
Statistical Analysis 1: Comparison: Placebo vs Reslizumab 110 mg; The frequency of CAEs was analyzed using the generalized linear model (GLM) for data from the negative binomial distributions that is commonly referred to as the negative binomial (NB) regression model. The primary NB model included the treatment group, randomization stratification factors, and number of prior exacerbations as model factors and the logarithm of treatment duration excluding the summed duration of exacerbations in the treatment period as an offset variable; Test type: Superiority — A fixed-sequence multiple testing procedure was implemented to test the primary and secondary endpoints while controlling the overall Type I error rate at 0.05. At the point where p>0.05, no further comparisons were interpreted inferentially; p = 0.194, Chi-squared — The treatment effect was tested using the likelihood based Chi-square test at the 0.05 significance level; CAE rate ratio (reslizumab vs placebo) = 0.79, 95% CI 2-sided [0.562 to 1.124]

2. Secondary Outcome: Change From Baseline to Week 52 in Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: Change in pre-bronchodilator FEV1 from baseline to week 52 is presented. FEV1 is a standard measurement of air movement in the lungs of participants with asthma obtained from pulmonary function tests. It is the volume of air expired in the first second of a forced expiration using a spirometer.
  Analysis of the change from baseline to each visit was performed using a mixed effect model for repeated measures (MMRM) including fixed effects for treatment, visit, treatment by visit interaction, age group, blood eosinophil counts at enrollment, and sex, height and baseline value as covariates, and participant as a random effect.
Time Frame: Baseline, Week 52
Population: ITT includes all randomized participants, excluding participants from the site terminated due to GCP issues. Treatment was based on the treatment to which participants were randomized, regardless of which treatment they received. Overall number of participants analyzed=participants with both baseline and Week 52 FEV1 values available.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 193 | 211
liters | 0.225 (0.040) | 0.368 (0.039)

3. Secondary Outcome: Change From Baseline to Week 52 in Asthma Quality of Life Questionnaire for Participants 12 Years and Older (AQLQ+12) Score
Description: AQLQ is a 32-item instrument administered as a self-assessment. AQLQ+12 is a modified version of AQLQ developed to measure functional impairments of participants aged 12-70 years. It is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Participants were asked to recall their experiences during the last 2 weeks and respond to each question on a 7-point scale (1=severe impairment, 7=no impairment), where higher scores indicated "better quality of life." Overall AQLQ+12 score is the mean of all 32 responses. Analysis of the change from baseline to each visit was performed using a MMRM including fixed effects for treatment, visit, treatment by visit interaction, age group, blood eosinophil counts at enrollment, and sex, height and baseline value as covariates, and participant as a random effect.
Time Frame: Baseline, Week 52
Population: Participants of the ITT population aged 12 to 70 years. Overall number of participants analyzed=participants with both baseline and Week 52 AQLQ+12 score available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 188 | 197
units on a scale | 1.06 (0.089) | 1.14 (0.087)

4. Secondary Outcome: Change From Baseline to Week 52 in 6-item Asthma Control Questionnaire (ACQ-6) Score
Description: The ACQ-6 is a 6-item validated asthma assessment tool that has been widely used. Six questions are self-assessments (completed by the participant), 5 questions assessing asthma symptoms: night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and 1 question for short-acting bronchodilator use. Each item on the ACQ-6 has a possible score ranges from 0 to 6, and the total score is the mean of all responses. The total score ranging from 0-6 (0=totally controlled and 6=severely uncontrolled). A higher score indicated poorer asthma control. Analysis of the change from baseline to each visit was performed using a mixed effect model for repeated measures (MMRM) including fixed effects for treatment, visit, treatment by visit interaction, age group, blood eosinophil counts at enrollment, and sex, height and baseline value as covariates, and participant as a random effect.
Time Frame: Baseline, Week 52
Population: ITT population includes all randomized participants, excluding those from the site terminated due to GCP issues. Treatment was based on the treatment to which participants were randomized, regardless of which treatment they received. Overall number of participants analyzed=participants with both baseline and Week 52 ACQ-6 score available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 197 | 212
units on a scale | -1.14 (0.080) | -1.22 (0.078)

5. Secondary Outcome: Change From Baseline to Week 52 in Total Asthma Symptom Scores (Day and Night)
Description: Asthma symptoms were recorded by participant each day and night in an asthma control diary. Night score was assessed on a 5-point scale where 0=no symptoms, slept through night, to 4=bad night, no sleep. Day score was assessed on a 6-point scale where 0=very well, no symptoms, to 5= asthma very severe, unable to carry out daily activities. Total asthma symptom score was calculated by taking the sum of the night and day asthma symptom scores recorded, ranging from 0 (no symptom) to 9 (severe symptom). A lower symptom score indicated a better outcome. Analysis of the change from baseline to each visit was performed using a MMRM including fixed effects for treatment, visit, treatment by visit interaction, age group, blood eosinophil counts at enrollment, and sex, height and baseline value as covariates, and participant as a random effect.
Time Frame: Baseline, Week 52
Population: ITT population included all randomized participants, excluding participants from site terminated due to GCP issues. Treatment was based on treatment to which participants were randomized, regardless of which treatment they received. Overall number of participants analyzed=participants with both baseline and Week 52 total asthma symptom score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 128 | 143
units on a scale | -1.4 (0.12) | -1.5 (0.12)

6. Secondary Outcome: Percentage of Asthma Control Days
Description: The percentage of asthma control days over 52 weeks of treatment is presented. An asthma control day was defined as a day on which the participant used less than or equal to 2 puffs of inhaled short-acting beta-agonist, had no nighttime awakenings, and experienced no asthma exacerbations. Analysis of the change from baseline to each visit was performed using a mixed effect MMRM including fixed effects for treatment, visit, treatment by visit interaction, age group, blood eosinophil counts at enrollment, and sex, height and baseline value as covariates, and participant as a random effect.
Time Frame: Day 1 to Week 52
Population: ITT population includes all randomized participants, excluding participants from the site terminated due to GCP issues. Treatment was based on the treatment to which participants were randomized, regardless of which treatment they actually received.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 230 | 234
percentage of days | 7.1 (1.27) | 8.0 (1.24)

7. Secondary Outcome: Change From Baseline to Week 32 in St. George's Respiratory Questionnaire (SGRQ) Total Score
Description: The SGRQ is a 17-item questionnaire with 50 weighted responses. It provides a total score and three component scores: Symptoms (distress caused by respiratory symptoms), Activity (physical activities that cause or are limited by breathlessness), and Impacts (social and psychological effects of the disease). The total score and each of the SGRQ subscores are scored from 0 to 100 where 0 indicates best and 100 indicates worst health. An increase in score indicates worsening health. Analysis of the change from baseline to each visit was performed using a mixed effect model for repeated measures (MMRM) including fixed effects for treatment, visit, treatment by visit interaction, age group, blood eosinophil counts at enrollment, and sex, height and baseline value as covariates, and participant as a random effect.
Time Frame: Baseline, Week 32
Population: ITT population includes all randomized participants, excluding participants from site terminated due to GCP issues. Treatment was based on treatment to which participants were randomized, regardless of which treatment they received. Overall number of participants analyzed= participants with both baseline and Week 32 SGRQ total scores available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 199 | 222
units on a scale | -13.1 (1.38) | -16.4 (1.32)

8. Secondary Outcome: Kaplan-Meier (K-M) Estimate of Probability (Percent [%]) of Not Experiencing a CAE by Week 52
Description: CAE was defined as a clinically judged deterioration in asthma control, as determined by the investigator and as evidenced by new or worsening asthma signs or symptoms based on the participant's history, asthma control diary, physical examination, and/or ambulatory or clinic visit assessment of lung function and that resulted in a medical intervention, including at least 1 of the following: 1) use of systemic corticosteroids (oral or injection) or at least a doubling from a stable maintenance oral corticosteroid dose for at least 3 days; 2) asthma-specific hospital admission; 3) asthma-specific emergency department visit.
  The KM method was used to estimate and compare the distributions of time to first CAE between treatment groups. Participants without an event during the treatment period were censored at either the date of the end of treatment (Week 52) visit for participants who completed treatment or at the date of last dose (+4 weeks) for participants who discontinued early.
Time Frame: Day 1 to Week 52
Population: ITT population includes all randomized participants, excluding participants from the site terminated due to GCP issues. Treatment was based on the treatment to which participants were randomized, regardless of which treatment they received.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 230 | 234
percent probability | 0.66 [0.59 to 0.72] | 0.66 [0.59 to 0.71]

9. Secondary Outcome: Number of CAEs Requiring Hospitalization and/or Emergency Department Visits During 52 Weeks of Treatment
Description: A CAE was defined as a clinically judged deterioration in asthma control, as determined by the investigator and as evidenced by new or worsening asthma signs or symptoms based on the participant's history, asthma control diary, physical examination, and/or ambulatory or clinic visit assessment of lung function and that resulted in a medical intervention, including at least 1 of the following: 1) use of systemic corticosteroids (oral or injection) or at least a doubling from a stable maintenance oral corticosteroid dose for at least 3 days; 2) asthma-specific hospital admission; 3) asthma-specific emergency department visit. The frequency of CAEs over 52-week treatment period is expressed as adjusted CAEs rate in 52 weeks. Adjusted CAE rate and confidence intervals were based on Negative Binomial regression model adjusted for stratification factors (age group, blood eosinophil group) and number of prior exacerbations, and an offset variable.
Time Frame: Day 1 to Week 52
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: events
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 230 | 234
events | 0.05 [0.016 to 0.169] | 0.05 [0.015 to 0.158]

10. Secondary Outcome: Number of Moderate Exacerbations During 52 Weeks of Treatment
Description: A moderate exacerbation was defined as a clinically judged deterioration in asthma control as determined by investigator and as evidenced by new or worsening asthma signs or symptoms based on the participant's history, asthma control diary, physical examination, and/or ambulatory or clinic visit assessment of lung function and that resulted in a medical intervention requiring additional asthma controller medication that was not a systemic corticosteroid and did not result in an asthma-specific hospitalization or emergency department visit (that is, a medical intervention that did not otherwise meet the criteria for primary endpoint). Frequency of moderate exacerbations over 52-week treatment period is expressed as adjusted exacerbation rate in 52 weeks. Adjusted exacerbation rate and confidence intervals were based on Negative Binomial regression model adjusted for stratification factors (age group, blood eosinophil group) and number of prior exacerbations, and an offset variable.
Time Frame: Day 1 to Week 52
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: events
Arm/Group | Placebo | Reslizumab 110 mg
Number analyzed (Participants) | 230 | 234
events | 0.15 [0.082 to 0.290] | 0.14 [0.074 to 0.250]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to the end of treatment visit (Week 52) for completed participants and between the first dose of study drug and 4 weeks after the last dose of study drug for participants who discontinued treatment early. Safety population includes all participants who received at least 1 dose of study drug (including from the site terminated due to GCP issues).
Description: 1 participant randomized to the placebo group was treated with reslizumab 110 mg at 1 study visit and counted in the reslizumab 110 mg arm for safety.There were no deaths during the treatment period. 1 death in the reslizumab group occurred 48 days after the participant's last dose.This participant's reason for discontinued was coded as death by the study site; but, the participant is not counted in all-cause mortality as the death occurred after the treatment period concluded.
Arm/Group | Placebo | Reslizumab 110 mg
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/237
Serious Adverse Events (participants affected / at risk) | 19/231 | 19/237
Other Adverse Events (participants affected / at risk) | 97/231 | 102/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=231) | Reslizumab 110 mg (N=237)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Reaction to food colouring (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign tracheal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis noninfective (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=231) | Reslizumab 110 mg (N=237)
Injection site erythema (General disorders) | 7 (13) | 13 (35)
Acute sinusitis (Infections and infestations) | 15 (19) | 14 (16)
Bronchitis (Infections and infestations) | 17 (23) | 13 (14)
Upper respiratory tract infection (Infections and infestations) | 19 (26) | 28 (37)
Viral upper respiratory tract infection (Infections and infestations) | 31 (42) | 27 (45)
Headache (Nervous system disorders) | 10 (19) | 14 (28)
Asthma (Respiratory, thoracic and mediastinal disorders) | 18 (25) | 9 (15)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT02452190/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT02452190/SAP_001.pdf